CLINICAL TRIAL: NCT05119595
Title: Prospective, Single Center PMCF-study on the Performance and Safety of the CranioFix®2 System Used for the Fixation of Craniotomized Bone Flaps and Fractures to the Neurocranium
Brief Title: PMCF Study on CranioFix®2 System Used for the Fixation of Craniotomized Bone Flaps and Fractures
Acronym: CRANFLAP
Status: Completed | Type: Observational
Sponsor: Aesculap AG (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-2043
Record Dates: First submitted 2021-10-07; First posted 2021-11-15 (Actual); Results first posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Skull Fractures
Keywords: Bone Flap Fixation; Fractures to the Neurocranium; Craniotomized bone flaps
MeSH Terms: conditions — Skull Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The CranioFix®2 PMCF study has been set up as an action within the framework of a proactive post-market surveillance system of the manufacturer. The aim of this observational study is to collect systematically and proactively data regarding the performance of CranioFix®2, like adverse events (AEs), handling and cosmetic outcome, under daily clinical practice when used as intended by the manufacturer.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age ≥ 18 years
* Use of CranioFix®2 system according to IfU
* Planned postoperative MRI within clinical routine

Exclusion Criteria:

* Pregnancy
* Patients with hypersensitivity to metals or allergies to the implant materials
* Inflammations in the region of the implant site
* Bone conditions that rule out the application of CranioFix®2 titanium clamps
* Use with artificial cranial bone flaps
* Bone tumors in the area supporting the implant
* Degenerative bone diseases
* Missing dura mater
* Application in the facial skull (viscerocranium) and in the orbital or skull-base region
* Combination of implant components from different manufacturers, i.e. additional use of plates and screws on the same bone fragment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients enrolled will be prospectively examined according to the study plan until follow-up examination (depending on routine in clinic).
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2022-03-22 (Actual); Primary Completion 2023-03-09 (Actual); Study Completion 2023-10-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Klinikum Stuttgart - Katharinenhospital, Stuttgart, Germany

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: CranioFix®2
Groups:
- Observational Study Group: All patients that were included in the study received treatment with the investigational device according to site's clinical routine.
Period: Overall Study
Arm/Group | Observational Study Group
Started (Due to a small defect size, only 2 clamps were used in 64% of cases. In 2 cases (8%), no indication was given as to how many CranioFix®2 clamps were used.) | 25; 53 CranioFix®2
Completed | 17; 33 CranioFix®2
Not Completed | 8; 20 CranioFix®2
Not completed — Death | 1
Not completed — Lost to Follow-up | 7

BASELINE CHARACTERISTICS:
Arm/Group | Observational Study Group
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Germany | 25

OUTCOME MEASURES:

1. Primary Outcome: Planarity of Bone Flap After Implantation
Description: The primary variable was the planarity of the bone flap after implantation. The bone flap planarity was evaluated as the rate of patients in which a dislocation of the bone flap occurred - defined as the height of the tilting (depression / protrusion) greater than the bone width.
Time Frame: Through postoperative course: at discharge (about up to 2 weeks after surgery) and post-operative follow-up (3±2 months after surgery)
Measure: Count of Participants; unit: Participants
Arm/Group | Observational Study Group
Number analyzed (Participants) | 25
Participants
  at discharge (about up to 2 weeks after surgery): yes | 23
  at discharge (about up to 2 weeks after surgery): no | 0
  at discharge (about up to 2 weeks after surgery): could not be evaluated | 2
  post-operative follow-up (3±2 months after surgery): yes | 17
  post-operative follow-up (3±2 months after surgery): no | 0
  post-operative follow-up (3±2 months after surgery): could not be evaluated | 8

2. Secondary Outcome: Number of Participants With Adverse Events (Intra- and Postoperative)
Description: Number of adverse events e.g. foreign body reactions, infections, injury to the dura, injury to the scalp, epiduralhaematoma, wound healing disorders with special focus on (serious) adverse events with (possible) relation to the investigational product
Time Frame: through study completion, an average of 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Observational Study Group
Number analyzed (Participants) | 25
Participants | 3

3. Secondary Outcome: Overall Handling of Instruments for CranioFix®2 System Implantation Documented on a Likert Scale
Description: Assessment of handling, documented on a Likert scale 1 to 5 (1 is the very good, 2 is good, 3 is acceptable, 4 is poor, 5 is very poor)
Time Frame: intraoperative
Measure: Number; unit: participants
Arm/Group | Observational Study Group
Number analyzed (Participants) | 25
participants
  very good | 12
  good | 12
  acceptable | 1
  poor | 0
  very poor | 0

4. Secondary Outcome: Stability of the Bone Flap After Fixation
Description: Assessment of stability of the bone flap, documented on a Likert scale 1 to 5 (1≙very good, 2≙good, 3≙medium, 4≙poor, 5≙very poor)
Time Frame: intraoperative, at discharge (about up to 2 weeks after surgery) and post-operative follow-up (3±2 months)
Population: One of 25 patients died after surgery before discharge, 7 patients were lost to follow-up between discharge and follow up visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Observational Study Group
Number analyzed (Participants) | 25
Participants
  surgery: very good | 19
  surgery: good | 5
  surgery: acceptable | 1
  surgery: could not be evaluated | 0
  at discharge: number analyzed (Participants) | 24
  at discharge: very good | 15
  at discharge: good | 8
  at discharge: acceptable | 0
  at discharge: could not be evaluated | 1
  at follow up (3±2 months: number analyzed (Participants) | 17
  at follow up (3±2 months: very good | 11
  at follow up (3±2 months: good | 6
  at follow up (3±2 months: acceptable | 0
  at follow up (3±2 months: could not be evaluated | 0

5. Secondary Outcome: Cosmetic Outcome
Description: Assessment of cosmetic outcome intraoperatively, at discharge and at post-operative follow-up documented on a 3 point scale (good, fair, bad)
Time Frame: intraoperative, at discharge (about up to 2 weeks after surgery) and post-operative follow-up (3±2 months)
Population: At the discharge visit, in 2 cases no evaluation of the cosmetic outcome by the surgeon was available because in one case no MRI scan was conducted and in another case the patient died after surgery before discharge.
  At the follow-up visit, in 8 cases, no evaluation of the cosmetic outcome was available because the follow-up visit did not take place.
Measure: Count of Participants; unit: Participants
Arm/Group | Observational Study Group
Number analyzed (Participants) | 25
Participants
  Cosmetic outcome by surgeon (surgery): good | 24
  Cosmetic outcome by surgeon (surgery): fair | 1
  Cosmetic outcome by surgeon (surgery): bad | 0
  Cosmetic outcome by surgeon (surgery): could not be evaluated | 0
  Cosmetic outcome by surgeon (discharge): number analyzed (Participants) | 24
  Cosmetic outcome by surgeon (discharge): good | 23
  Cosmetic outcome by surgeon (discharge): fair | 0
  Cosmetic outcome by surgeon (discharge): bad | 0
  Cosmetic outcome by surgeon (discharge): could not be evaluated | 1
  Cosmetic outcome by surgeon (follow up): number analyzed (Participants) | 17
  Cosmetic outcome by surgeon (follow up): good | 17
  Cosmetic outcome by surgeon (follow up): fair | 0
  Cosmetic outcome by surgeon (follow up): bad | 0
  Cosmetic outcome by surgeon (follow up): could not be evaluated | 0
  Cosmetic outcome by patient (discharge): number analyzed (Participants) | 24
  Cosmetic outcome by patient (discharge): good | 22
  Cosmetic outcome by patient (discharge): fair | 1
  Cosmetic outcome by patient (discharge): bad | 0
  Cosmetic outcome by patient (discharge): could not be evaluated | 1
  Cosmetic outcome by patient (follow up): number analyzed (Participants) | 17
  Cosmetic outcome by patient (follow up): good | 14
  Cosmetic outcome by patient (follow up): fair | 3
  Cosmetic outcome by patient (follow up): bad | 0
  Cosmetic outcome by patient (follow up): could not be evaluated | 0

ADVERSE EVENTS:
Time Frame: 3 ± 2 months
Groups:
- Observational Study Group: In total, 3 adverse events were reported in 3 study patients. Two of the three AEs were classified as serious adverse events.
  In 2 of the AEs a measure was taken which included non-operative measures (n = 1) and reoperation (n = 1), in 1 of the AE no therapeutic measure due to the AE was taken (n=1). No causal relationship to the investigational device was stated in any of the cases. Consequently, none of the AE is related to be an ADE (Adverse Device Effect).
Arm/Group | Observational Study Group
All-Cause Mortality (participants affected / at risk) | 1/25
Serious Adverse Events (participants affected / at risk) | 2/25
Other Adverse Events (participants affected / at risk) | 1/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Observational Study Group (N=25)
Intracerebral hemorrhage after resection with generalized seizure and hemiparesis on the right side. (Injury, poisoning and procedural complications) | 1 (1) — Probably the hemorrhage was caused by occlusion of the draining veine.
Intracerebral hemorrhage after resection (Injury, poisoning and procedural complications) | 1 (1) — Probably the bleeding was caused by the tumor resection.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Observational Study Group (N=25)
Epidural collection of liquid and air in access area, non-space-consuming.Clinically inapparent. (Injury, poisoning and procedural complications) | 1 (1) — Extension of epidural space might be caused by large defect of brain

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The clinic will ensure that a manuscript intended for publication that is related to this study is made available to the sponsor for review before submission in order to give the sponsor the opportunity to comment. Furthermore, the clinic ensures that an abstract intended for presentation, as well as a manuscript intended for this purpose and the presentation slides themselves, are sent to the sponsor before submission to a congress.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-09-24): https://cdn.clinicaltrials.gov/large-docs/95/NCT05119595/Prot_SAP_000.pdf